CLINICAL TRIAL: NCT07087704
Title: Effects of a Chilean Diet Supplemented With Gevuina Avellana on Lipid Profile in Humans With Hypercholesterolemia
Acronym: PRODICHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Concepcion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBB 530-2019-M; CEC-SSC: 21-09-48 (Other: Comité Ético Científico del Servicio de Salud Concepción); ANID FONDECYT INICIACION (Other: 1119064)
Record Dates: First submitted 2025-07-09; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Hypercholesterolemia
Keywords: lipid profile; chilean diet; Gevuina avellana; Cardiovascular disease prevention; nutritional intervention; chilean hazelnut
MeSH Terms: conditions — Hypercholesterolemia | interventions — Diet, High-Fat; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-fat diet (Active Comparator): The control group maintained a low-fat diet (<30% total energy value) based on the Ministerio de Salud de Chile (MINSAL) technical guidelines for dyslipidemia management
  Interventions: Dietary Supplement: Low-fat diet
- High-fat Chilean diet supplemented with Gevuina avellana (Experimental): The experimental group followed a Chilean diet (adapted from the Mediterranean Diet using Chilean ingredients) supplemented with 30 g/day of Gevuina avellana and a diet of 40% total energy value
  Interventions: Dietary Supplement: High-fat diet

INTERVENTIONS:
Dietary Supplement: High-fat diet — The group follows a Chilean diet (adapted from the Mediterranean Diet using Chilean ingredients) supplemented with 30 g/day of Gevuina avellana and providing 40% of total energy value from fat. To promote adherence to the diet, individual motivational interviews and group sessions (with approximately 25 participants) are conducted once per month. Each participant is provided once a month with individually packaged Chilean hazelnuts to reach a daily intake of 30 g.
  Other Names: Chilean hazelnut supplementation; Gevuina avellana supplementation
  Arms: High-fat Chilean diet supplemented with Gevuina avellana
Dietary Supplement: Low-fat diet — The group maintains a low-fat diet (<30% of total energy value) based on the Chilean Ministry of Health (MINSAL) technical guidelines for dyslipidemia management. To promote adherence to the diet, individual motivational interviews and group sessions (with approximately 25 participants) are conducted once per month.
  Other Names: MINSAL guidelines for dyslipidemia management; Chilean Ministry of Health technical guidelines for dyslipidemia management
  Arms: Low-fat diet

SUMMARY:
The purpose of this study is to determine if supplementing a Chilean diet with Chilean hazelnut (Gevuina avellana) improves cholesterol levels in adults with hypercholesterolemia. The main question is whether this supplementation reduces total serum cholesterol compared to a low-fat diet without hazelnut.

DETAILED DESCRIPTION:
This is a 6-month randomized controlled parallel study involving hypercholesterolemic volunteers (serum cholesterol > 200 mg/dL, with or without triglycerides > 150 mg/dL) aged 18-60 years from Concepción, Chile. Participants are randomly assigned to two groups:

Intervention group: Receives the Chilean diet supplemented daily with 30 g of Chilean hazelnut (Gevuina avellana).

Control group: Receives dietary advice to follow a low-fat diet based on American Heart Association recommendations, without hazelnut supplementation.

Primary outcome is total serum cholesterol. Secondary assessments include anthropometric measures, blood pressure, diet adherence, physical activity, sociodemographic variables, smoking habits, medical diagnoses, medication use, and biochemical markers of lipid profile, oxidative damage, antioxidant capacity, endothelial peptides, and inflammation.

Data collection occurs at baseline, 2, 4, and 6 months. Individual motivational interviews and group motivational sessions (approximately 25 participants each) are conducted to enhance adherence. Blood samples for lipid profiling and other biochemical analyses are collected fasting at baseline and study completion.

Blood fractionation is performed to obtain plasma, serum, erythrocytes, and peripheral blood mononuclear cells (PBMCs) for detailed fatty acid profiling and biomarker measurements.

This study aims to provide insight into the potential cardiovascular benefits of Gevuina avellana supplementation in a Chilean dietary context.

ELIGIBILITY:
Inclusion Criteria:

* Serum cholesterol level greater than 200 mg/dL with or without triacylglycerol greater than 150 mg/dL
* Have received both doses included in the SARS-CoV-2 vaccination campaign and possess their corresponding mobility pass.

Exclusion Criteria:

* Be undergoing medical treatment for hypercholesterolemia.
* Have systemic diseases such as diabetes, hypertension, kidney, or liver disease.
* Pregnant or breastfeeding women.
* Have a household member or close relative who has been previously recruited.
* Have allergies to tree nuts.
* Have an electronic implant such as a pacemaker.
* Also, individuals who do not meet the minimum conditions compatible with the study modality will not be able to participate in the intervention, such as: having access to an electronic device such as a cellphone or computer; having access to mobile internet or Wi-Fi at home; or having the necessary knowledge or support to use the platform

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Total cholesterol (mg/dL) | From enrollment to the end of treatment at 6 months
  Total serum cholesterol under fasting condition

SECONDARY OUTCOMES:
Blood pressure (mmHg) | From enrollment to the end of treatment at 6 months
  Blood pressure measured by a semi-automatic sphygmomanometer
Body weight (kg) | From enrollment to the end of treatment at 6 months
  Body weight is measured using a portable digital scale (Seca®) with a precision of 100 g, placed on a flat, horizontal, and firm surface. Participants are asked to remove their shoes and wear minimal clothing to ensure accurate measurement.
Height (m) | From enrollment to the end of treatment at 6 months
  Height is measured using a portable stadiometer (Seca® 213) with 0.1 cm precision. Participants stand barefoot with heels together (forming a 45-60° angle), back straight and in contact with the stadiometer, fully extended. The head is positioned in the Frankfurt horizontal plane. Participants are instructed to take a deep breath and remain still. The headpiece is gently lowered to contact the head, applying slight pressure to compress the hair.
Body Mass Index (kg/m2) | From enrollment to the end of treatment at 6 months
  Weight and height will be combined to report BMI in kg/m2)
Waist circumference (mm) | From enrollment to the end of treatment at 6 months
  Waist circumference is measured using a non-stretchable measuring tape (Seca® 201) with 0.1 cm precision. The participant stands upright, shirtless or with the waist area exposed, feet 25-30 cm apart, arms relaxed at the sides, and weight evenly distributed. Measurement is taken at the midpoint between the lower rib and the iliac crest along the midaxillary line. Reference points are palpated and marked. The tape is placed horizontally, snug but not compressing soft tissues, and measurement is taken at the end of a normal exhalation. Two measurements are taken; if they differ by more than 1 cm, a third is taken. The final value is the average of the two closest readings.
LDL cholesterol (mg/dL) | From enrollment to the end of treatment at 6 months
  LDL cholesterol under fasting condition
HDL cholesterol (mg/dL) | From enrollment to the end of treatment at 6 months
  HDL cholesterol under fasting condition
Triglycerides (mg/dL) | From enrollment to the end of treatment at 6 months
  Triglycerides under fasting condition
Superoxide dismutase activity | From enrollment to the end of treatment at 6 months
  Superoxide dismutase activity is measured in plasma and erythrocytes using spectrophotometric methods.
Catalase activity | From enrollment to the end of treatment at 6 months
  Catalase is measured in plasma and erythrocytes using spectrophotometric methods.
Homocysteine | From enrollment to the end of treatment at 6 months
  Plasma homocysteine is measured using a commercial ELISA kit, following the manufacturer's instructions.
Adiponectin | From enrollment to the end of treatment at 6 months
  Adiponectin levels in plasma are measured using a commercial ELISA kit according to the manufacturer's protocol
Oxidized low-density lipoprotein (LDLox) | From enrollment to the end of treatment at 6 months
  Oxidized low-density lipoprotein (LDLox) levels in plasma are measured using a commercial ELISA kit following the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Martorell, PhD, Principal Investigator — Centro de Vida Saludable
Locations (1):
- Laboratorio Prevegen, Concepción, Región del Biobío, Chile

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, ICF
Time Frame: Once the results are published
Access Criteria: Contact to Miquel Martorell at mmartorell@udec.cl Explain the data required and the purpose of use

REFERENCES:
- See also: Research Thesis on Plasma Biochemical Markers — https://vidasaludable.udec.cl/node/918
- See also: Research Thesis on PBMCs Biochemical Markers — https://vidasaludable.udec.cl/node/573